CLINICAL TRIAL: NCT01462266
Title: A Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Study the Safety and Insulin-Sparing Efficacy of the Addition of Sitagliptin in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Insulin Alone or in Combination With Metformin
Brief Title: Study of Sitagliptin for the Treatment of Type 2 Diabetes Mellitus With Inadequate Glycemic Control on Insulin (MK-0431-260)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-260
Record Dates: First submitted 2011-10-27; First posted 2011-10-31 (Estimated); Results first posted 2014-04-08 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Insulin Glargine; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin (Experimental): Sitagliptin 100 mg once daily
  Interventions: Drug: Sitagliptin; Biological: Insulin Glargine; Drug: Metformin
- Placebo (Placebo Comparator): Placebo to sitagliptin once daily
  Interventions: Drug: Comparator: Placebo; Biological: Insulin Glargine; Drug: Metformin

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin 100 mg tablet once daily for 24 weeks
  Other Names: Januvia
  Arms: Sitagliptin
Drug: Comparator: Placebo — Placebo to sitagliptin once daily for 24 weeks
  Arms: Placebo
Biological: Insulin Glargine — Participants on insulin glargine or another insulin regimen for at least 10 weeks prior to screening will continue or switch to open-label insulin glargine once-daily in the evening for the duration of the study.
Drug: Metformin — Participants on metformin oral tablet(s) at a dose of at least 1500 mg/day for at least 10 weeks prior to screening will continue receiving metformin at their current dose for the duration of the study.
  Other Names: Glucophage

SUMMARY:
The purpose of this study is to examine the insulin-sparing effect of sitagliptin 100 mg once-daily compared with placebo over 24 weeks in participants with type 2 diabetes mellitus who have inadequate glycemic control on insulin alone or in combination with metformin. The primary hypothesis of this study is that after 24 weeks, sitagliptin reduces the dose of insulin relative to placebo.

ELIGIBILITY:
Inclusion Criteria:

* has type 2 diabetes mellitus
* has one of the following criteria:

  * diagnosed with diabetes after age 40 years and insulin therapy was initiated at least 3 years following diagnosis
  * if diagnosed with diabetes under age 40 years or insulin started earlier than 3 years after diagnosis, has a fasting C-peptide greater than 0.7 ng/mL
* must be at least 18 years of age and less than or equal to 80 years of age (for participants in India: must be at least 18 years of age and less than or equal to 65 years of age)
* on a stable regimen of insulin for at least 10 weeks with or without metformin (at least 1500 mg/day) and/or sulfonylurea for at least 10 weeks
* is highly unlikely to become pregnant (not of reproductive potential or agrees to remain abstinent or use (or have their partner use) an acceptable method of birth control during the study and for 14 days after the last dose of study medication

Exclusion Criteria:

* has been treated with a dipeptidyl peptidase IV (DPP-4) inhibitor, a thiazolidinedione (TZD), or a glucagon-like peptide-1 (GLP-1) mimetic or analogue, within the past 12 weeks
* currently on treatment with daily use (one or more injections per day) of a

pre-prandial short-acting or rapid-acting insulin alone or as part of a basal/bolus insulin regimen

* has symptomatic hyperglycemia that requires immediate initiation, adjustment, or addition of antihyperglycemic therapy
* has a history of 2 or more episodes of hypoglycemia resulting in seizure,

coma, or loss of consciousness, - or - has had recurrent (≥3 times per week) episodes of hypoglycemia over the past 8 weeks

* has a history of ketoacidosis
* is not appropriate for or does not agree to target a fasting glucose of 72-100 mg/dL [4.0-5.6 mmol/L]
* is on or likely to require treatment with corticosteroids
* has undergone a surgical procedure within 4 weeks or has planned major surgery during the study
* is currently being treated for hyperthyroidism or is on thyroid hormone

therapy and has not been on a stable dose for at least 6 weeks

* has a history of active liver disease (other than non-alcoholic hepatic

steatosis)

* has had new or worsening signs or symptoms of coronary heart disease or

congestive heart failure within the past 3 months, or has any of the following

disorders within the past 3 months:

* acute coronary syndrome
* coronary artery intervention
* stroke or transient ischemic neurological disorder

  * has a systolic blood pressure greater than 160 mm Hg or a diastolic blood pressure greater than 90 mm Hg
  * has human immunodeficiency virus (HIV)
  * has severe peripheral vascular disease
  * has a clinically important hematological disorder
  * has a history of malignancy that is less than 5 years from study start, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer
  * has a positive urine pregnancy test
  * is pregnant or breast-feeding, or is expecting to conceive or donate eggs

during the study

* a user of recreational or illicit drugs or has had a recent history of drug abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2012-01-13 (Actual); Primary Completion 2013-06-06 (Actual); Study Completion 2013-06-07 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Mathieu C, Shankar RR, Lorber D, Umpierrez G, Wu F, Xu L, Golm GT, Latham M, Kaufman KD, Engel SS. A Randomized Clinical Trial to Evaluate the Efficacy and Safety of Co-Administration of Sitagliptin with Intensively Titrated Insulin Glargine. Diabetes Ther. 2015 Jun;6(2):127-42. doi: 10.1007/s13300-015-0105-3. Epub 2015 Mar 28. PMID 25820927
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0431-260&kw=0431-260&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Sitagliptin: Sitagliptin 100 mg administered orally once daily for 24 weeks.
- Placebo: Placebo to sitagliptin administered orally once daily for 24 weeks.
Period: Overall Study
Arm/Group | Sitagliptin | Placebo
Started | 330 | 330
Treated | 329 (One participant was randomized in error and did not receive study medication.) | 329 (One participant was randomized in error and did not receive study medication.)
Completed | 295 | 303
Not Completed | 35 | 27
Not completed — Adverse Event | 7 | 6
Not completed — Death | 2 | 1
Not completed — Lack of Efficacy | 0 | 2
Not completed — Lost to Follow-up | 4 | 3
Not completed — Non-compliance with study drug | 3 | 0
Not completed — Creatinine and eGFR, excluded medication | 8 | 4
Not completed — Physician Decision | 2 | 5
Not completed — Protocol Violation | 1 | 3
Not completed — Withdrawal by Subject | 7 | 2
Not completed — Screen failure | 1 | 1

BASELINE CHARACTERISTICS:
Population: One participant in both the Sitagliptin group and Placebo group was randomized in error and did not receive study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Placebo | Total
Number analyzed (Participants) | 329 | 329 | 658
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.3 (8.9) | 58.3 (9.7) | 58.8 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178 | 165 | 343
  Male | 151 | 164 | 315

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Daily Insulin Dose at Week 24
Description: Change in daily insulin dose following 24 weeks of therapy (i.e., daily insulin dose at Week 24 minus daily insulin dose at baseline)
Time Frame: Baseline and Week 24
Population: Full Analysis Set (FAS) population included all randomized participants who took at least one dose of study medication and had at least one measurement either at baseline or post-randomization.
Measure: Least Squares Mean (95% Confidence Interval); unit: International Units (IU)
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 329 | 329
International Units (IU) | 19.0 (19.6) [16.5 to 21.6] | 23.8 (24.0) [21.3 to 26.3]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p = 0.009, Longitudinal data analysis; Adjusting for participant's use of metformin at Visit 1/Screening Visit (i.e., on metformin, or not on metformin); Mean Difference (Final Values) = -4.7, 95% CI 2-sided [-8.3 to -1.2]

2. Secondary Outcome: Change From Baseline in Hemoglobin A1c (A1C) at Week 24
Description: A1C is measured as the percentage of glycosylated hemoglobin. Change in A1C following 24 weeks of therapy (i.e., A1C at Week 24 minus A1C at baseline)
Time Frame: Baseline and Week 24
Population: FAS population included all randomized participants who took at least one dose of study medication and had at least one measurement either at baseline or post-randomization.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent of total hemoglobin
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 329 | 329
Percent of total hemoglobin | -1.31 (0.98) [-1.43 to -1.20] | -0.87 (1.10) [-0.98 to -0.75]

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: Change in FPG (before breakfast) following 24 weeks of therapy (i.e., FPG at Week 24 minus FPG at baseline)
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 329 | 329
mg/dL | -55.5 (52.0) [-61.1 to -49.9] | -44.8 (62.4) [-50.4 to -39.2]

4. Secondary Outcome: Percent of Participants Achieving Fasting Glucose Target at Any Time During the Study
Description: The fasting glucose target was defined as 3 consecutive days with a fingerstick glucose of 72 to 100 mg/dL (4.0 - 5.6 mmol/L).
Time Frame: Up to 24 weeks
Population: FAS population included all randomized participants who took at least one dose of study medication, and had at least one post-randomization glycemic goal assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 327 | 326
Percentage of participants | 77.4 [72.6 to 82.2] | 74.1 [69.0 to 79.2]

5. Secondary Outcome: Time to Achieve the Fasting Glucose Target
Description: Fasting glucose target 3 consecutive days with a fingerstick glucose of 72 to 100 mg/dL (4.0 - 5.6 mmol/L). This analysis was the Kaplan-Meier estimated 50th percentile of time (days) to first attainment of target.
Time Frame: Up to 24 weeks
Population: FAS population included all randomized participants who took at least one dose of study medication and had at least one post-randomization glycemic goal assessment.
Measure: Median (95% Confidence Interval); unit: Days to first attainment of target
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 253 | 242
Days to first attainment of target | 78 [64 to 85] | 90 [80 to 107]

ADVERSE EVENTS:
Time Frame: Up to Week 24 + 14-day follow-up
Arm/Group | Sitagliptin | Placebo
Serious Adverse Events (participants affected / at risk) | 13/329 | 12/329
Other Adverse Events (participants affected / at risk) | 121/329 | 168/329
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=329) | Placebo (N=329)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Spermatocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=329) | Placebo (N=329)
Diarrhoea (Gastrointestinal disorders) | 17 (19) | 11 (11)
Nasopharyngitis (Infections and infestations) | 13 (16) | 26 (29)
Urinary tract infection (Infections and infestations) | 14 (16) | 17 (18)
Hypoglycaemia (Metabolism and nutrition disorders) | 93 (358) | 144 (794)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.